CLINICAL TRIAL: NCT00157560
Title: A Phase II Trial of ModifiedTriple Doublet Therapy in the Treatment of Women With Newly Diagnosed Carcinoma of Müllerian Origin
Brief Title: Phase II Study of Modified Triple Doublet Therapy in Women With Newly Diagnosed Mullerian Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: GlaxoSmithKline (Industry); Eli Lilly and Company (Industry)
Responsible Party: Maria Roche, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00-305
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2008-01-03 (Estimated); Status verified 2007-12

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Chemotherapy, multiple agents

SUMMARY:
Over the last few years several novel agents have been defined which are active in the treatment of relapsed epithelial ovarian carcinoma. Many of these new agents seemed to have mechanisms of action that are different from Carboplatin and taxol. This trial looks to evaluate the effectiveness and toxicity of three sequential chemotherapy doublets in the treatment of women with newly diagnosed ovarian, primary peritoneal or tubal carcinoma.

DETAILED DESCRIPTION:
Objective: To evaluate a novel regimen in ovarian carcinoma with an aim of demonstrating a higher than 50% laparotomy defined response rate. This rate is defined as the proportion of patients achieving either a pathologic complete response or a microscopic positive second look at the conclusion of therapy.

Primary study goals:

· To determine the efficacy of a triple doublet regimen in carefully defined cohorts of patients as defined by the surgical defined response rate

Secondary study goals:

* To evaluate incidence of tubulin mutations in primary and secondary surgical specimens.
* To evaluate changes in IL-6, IL-8, VEGF, and FGF, at primary diagnosis, during and at the conclusion of therapy.
* To describe initial IL-6, IL-8, and FGF levels in patients who ultimately achieve pathologic remission vs those with gross residual disease.

Patients will recieve 3 cycles of carboplatin and gemcitabine followed by 3 cycles of taxol and carboplatin and then three cycles of adriamycin and topotecan. All patients with a clinically complete response will then undergo second look operation to determine pathologically defined response.

* SLO = Second Look Operation

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed epithelial carcinoma of müllerian origin. Specifically, ovarian, primary peritoneal and tubal carcinoma will be allowed. All histologic subtypes are eligible.

  * Patients must have undergone an attempt at aggressive surgical debulking or alternatively be eligible for interim debulking after cycle #3. Patients debulked to no evidence of disease, microscopic disease or gross residual disease are eligible.
  * Stage II, III or IV disease. Patients with disease outside the abdominal cavity are eligible unless presentation includes brain metastases.
  * Able and willing to undergo a second look staging laparotomy.
  * Patients must give written informed consent.
  * Patient must be ag· Performance status (ECOG) >2.
  * Previous chemotherapy.
  * Creatinine > 1.5
  * History of recent MI or congestive heart failure within 6 months of surgery
  * SGOT > 2x ULN, bilirubin > 1.5 X ULN
  * Concurrent invasive malignancy. (Patients with concurrent superficial endometrial carcinoma are eligible if their endometrial carcinoma is superficial or invades less than 50% the thickness of the myometrium).
  * Known hypersensitivity to E.coli derived products?
  * Active psychiatric or mental illness that makes informed consent or careful clinical follow-up unlikely e 18 years or older.
  * Adequate bone marrow function with an ANC > 2,500 and Platelets >100,000/mm3.

Exclusion Criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83
Dates: Start 2000-12; Primary Completion 2006-11 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
· To determine the efficacy of the triple doublet regimen as defined by second look laparotomy

SECONDARY OUTCOMES:
· To evaluate incidence of tubulin mutations in primary and secondary surgical specimens.
· To evaluate changes in IL-6, IL-8, VEGF, and FGF at primary diagnosis, during and at the conclusion of therapy.
· To describe initial IL-6 levels in patients who ultimately achieve pathologic remission vs those with gross residual disease at the time of SLO.

CONTACTS AND LOCATIONS:
Overall Officials: Michael V Seiden, M.D. Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: Related Info — http://www.dfhcc.org